CLINICAL TRIAL: NCT05220423
Title: Impact of an SMS Reminder on Influenza Vaccination Coverage in Patients With Rheumatoid Arthritis Taking Anti-TNF : an Ancillary Study to the French National Registry ART E-cohort
Brief Title: Effectiveness of SMS Reminders on Influenza Vaccination Coverage in Patients With RA in the ART Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Societe Francaise de Rhumatologie (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ART- Influenza
Record Dates: First submitted 2021-12-23; First posted 2022-02-02 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis
Keywords: anti-TNF; Flu; influenza; vaccination; biologics; bDMARDs; targeted therapies
MeSH Terms: conditions — Arthritis, Rheumatoid; Influenza, Human | interventions — Spermine Synthase

STUDY DESIGN:
Who Masked: Participant
Masking Description: patient reported outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminders Group (Other): This group will receive 6 reminders (sms/emails) on top of the National annual communication campaign organized by the French Health System authorities
  Interventions: Other: sms and emails reminders
- No reminders group (Other): This group will receive no reminders on top of the National annual communication campaign organized by the French Health System authorities
  Interventions: Other: No reminders

INTERVENTIONS:
Other: sms and emails reminders — 6 reminders encouraging influenza vaccination on top of the National annual communication campaign organized by the French Health System authorities
  Arms: Reminders Group
Other: No reminders — no reminders on top of the National annual communication campaign organized by the French Health System authorities
  Arms: No reminders group

SUMMARY:
Biotherapies have significantly improved the prognosis of rheumatoid arthritis (RA), particularly anti-TNF. However, these molecules are associated with a well-demonstrated increase in infectious risk, including an over-risk of pneumococcal and influenza infection.. Therefore, when initiating anti-TNF treatments, it is recommended to update the vaccination schedule of these patients, to vaccinate them against pneumococcus and carry out an annual anti influenza vaccination.. However, vaccination coverage remains sub-optimal. The means to improve this vaccination coverage are multiple but often require human resources. Medical teams often lack time, nursing interventions are effective but again requires the availability of the health care team. The use of modern digital means (automatic reminders) is an attractive alternative to increase immunization coverage without the use of medical or paramedical time.

The objective of the study is to evaluate the effectiveness, in terms of immunization coverage, of SMS and/or email reminders reminding the need to vaccinate against seasonal influenza compared to usual care, in patients with RA on biotherapies participating in the e-cohort of the French ART Registry (NCT03062865).

This study will be based on the ART Registry e-cohort. This will be a randomized controlled trial in patients in the ART e-cohort. The patients will be allocated in one of the 2 arms : one arm receiving reminders by email and SMS of the influenza vaccination, the other arm with absence of reminders. This study will be conducted during the annual French National communication campaign to encourage influenza vaccination.

The main evaluation criterion will be the influenza vaccination coverage rate at the end of the vaccination campaign. It will be compared between the two arms.

DETAILED DESCRIPTION:
Design :

Randomised, controlled trial within the e-cohort population of the French ART registry (observational study)

Target population :

All participants to the e-cohort of the French ART Registry (Rheumatoid Arthritis and anti-TNF)

ELIGIBILITY:
All patients included in the French ART Registry (rheumatoid arthritis and anti-TNF) and participating to the e-cohort.

Inclusion Criteria:

* Adult patients with RA,
* Patient in whom the specialist physician decides to start treatment with an anti-TNF drug, regardless of the treatment line and regardless of the anti-TNF, including infliximab, adalimumab, etanercept, certolizumab and golimumab, and their respective biosimilar according to their arrival on the market
* Clinicians (hospital-based and private practice) who agree to adhere to the yearly renewal of the hospital prescription

Exclusion Criteria:

* Patient already treated by the same anti-TNF in the past (same drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Influenza vaccination coverage | up to 5 months
  The vaccination coverage will be evaluated by comparing the vaccination coverage rate between both groups

SECONDARY OUTCOMES:
Influenza vaccination coverage in the non-intervention group post Covid 19 pandemia | up to 5 months
  Comparison of the actual vaccination rate with the 2019-2020 vaccination rate
Factors associated with influenza non-vaccination | up to 5 months
  identification of the factors associated with the absence of vaccination assessed by questionnaire
Reasons for influenza vaccination and non-vaccination | up to 5 months
  Number of patients for each reason for vaccination and non-vaccination assessed by questionnaire
Covid-19 vaccination coverage including primo vaccination, booster | up to 5 months
  Estimation of the actual covid19 vaccination coverage rate
Adherence to national recommendations on COVID vaccination in patients with immunosuppressive treatment | up to 5 months
  Estimation of the actual covid19 vaccination coverage rate in patients with immunosuppressive treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raphaele Seror, Principal Investigator — Hôpital Bicêtre; Adeline Ruyssen-Witrand, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen Y, Baron G, Hamamouche N, Belkhir R, Miconnet S, Soubrier M, Hostachy C, Thevenot P, Basch A, Truchetet ME, Claudepierre P, Dernis E, Marotte H, Flipo RM, Brocq O, Morel J, Fautrel B, Salliot C, Saraux A, Leske C, Schaeverbeke T, Ravaud P, Mariette X, Ruyssen-Witrand A, Seror R; ART Study Group section sign. Do SMS/e-mail reminders increase influenza vaccination of rheumatoid arthritis patients under anti-TNF: a nested randomized controlled trial in the ART e-cohort. Rheumatology (Oxford). 2025 May 1;64(5):2496-2504. doi: 10.1093/rheumatology/keae599. PMID 39576675
- See also: French National Registry - ART — https://clinicaltrials.gov/ct2/show/NCT03062865